CLINICAL TRIAL: NCT05157243
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Efficacy and Safety of Nitazoxanide for Treatment of Mild or Moderate COVID-19 in Subjects at High Risk of Severe Illness
Brief Title: Trial to Evaluate Nitazoxanide for Treatment of Mild or Moderate COVID-19 in Subjects at High Risk of Severe Illness
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM08-3010
Record Dates: First submitted 2021-12-10; First posted 2021-12-14 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide; Standard of Care

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized 1:1 to receive 600mg NTZ or placebo twice daily for 5 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Experimental): Nitazoxanide 300 mg extended release tablets
  Interventions: Drug: Nitazoxanide; Dietary Supplement: Vitamin Super-B Complex; Other: Standard of Care
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Dietary Supplement: Vitamin Super-B Complex; Drug: Placebo; Other: Standard of Care

INTERVENTIONS:
Drug: Nitazoxanide — Two NTZ 300 mg extended release tablets administered orally with food twice daily for 5 days
  Other Names: NTZ; NT-300
  Arms: Nitazoxanide
Dietary Supplement: Vitamin Super-B Complex — Vitamin Super B-Complex administered orally twice daily for 5 days to maintain the blind
Drug: Placebo — Two matching placebo tablets administered orally with food twice daily for 5 days
  Arms: Placebo
Other: Standard of Care — Local standard of care for COVID-19
  Other Names: SOC

SUMMARY:
The purpose of this study is to determine whether nitazoxanide (NTZ) is safe and effective in treating mild or moderate COVID-19 illness in adults and adolescents at highest risk for severe outcomes. Each participant will be followed for approximately 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 12 years of age
* At high risk of progressing to severe COVID-19 illness due to having one of the following underlying conditions and/or sociodemographic risk factors:

  1. Age ≥ 55 years (with or without comorbidities),
  2. Body mass index (BMI) ≥30 kg/m² if ≥ 18 years of age or BMI ≥85th percentile for age and gender based on CDC growth charts,
  3. Chronic kidney disease,
  4. Diabetes,
  5. Immunosuppressive disease,
  6. Currently receiving immunosuppressive treatment,
  7. Cardiovascular disease (including congenital heart disease) or hypertension,
  8. Chronic lung disease (e.g., chronic obstructive pulmonary disease, moderate-to-severe asthma, interstitial lung disease, cystic fibrosis, pulmonary hypertension),
  9. Sickle cell disease,
  10. Neurodevelopmental disorders or other conditions that confer medical complexity.
* Positive test for SARS-CoV-2 by RT-PCR or validated rapid antigen test within 72 hours prior to enrollment in the trial (positive sample must be collected within 72 hours prior to enrollment).
* Presence of symptoms consistent with mild or moderate COVID-19 in the judgment of the Investigator.
* Onset of symptoms no more than 72 hours before enrollment in the trial. Onset of symptoms is defined as the earlier of the first time at which the subject experienced subjective fever or any respiratory symptom (headache/head congestion, throat symptoms, nasal symptoms, chest symptoms, cough).
* Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of all protocol procedures.

Exclusion Criteria:

* Persons with any clinical signs or symptoms suggestive of severe systemic illness with COVID-19, including the following:

  1. shortness of breath at rest
  2. resting pulse ≥125 beats per minute
  3. resting respiratory rate ≥30 breaths per minute
  4. Oxygen saturation ≤ 93% on room air at sea level
* Immunocompetent persons who have been fully vaccinated for SARS-CoV-2, defined as having received all expected vaccine doses for a 2-dose or single-dose series at least two weeks prior to onset of symptoms.
* Females of childbearing potential who are either pregnant or sexually active without the use of birth control.
* Subjects residing in the same household with another subject participating in the study.
* Treatment with any investigational drug or vaccine therapy within 30 days prior to screening.
* Receipt of monoclonal antibody therapy for COVID-19 within the preceding 90 days.
* Receipt of any dose of NTZ within seven days prior to screening.
* Known sensitivity to NTZ or any of the excipients comprising the study medication.
* Subjects unable to swallow oral tablets or capsules.
* Subjects with known severe heart, lung, neurological or other systemic disease that the Investigator believes could preclude safe participation.
* Subjects likely or expected to require hospitalization unrelated to COVID-19 during the study period.
* Subjects taking medications considered to be major CYP2C8 substrates.
* Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants progressing to severe COVID-19 or death from any cause | Day 1 through Day 28

OTHER OUTCOMES:
Proportion of participants with COVID-19-related hospitalization or death from any cause | Day 1 through Day 28
Change in cytokine levels | Day 1 through Day 4